CLINICAL TRIAL: NCT04228432
Title: E-monitoring of Patients Under Adjuvant Hormonotherapy for Breast Cancer: Pilot Study
Brief Title: E-monitoring of Patients Under Adjuvant Hormonotherapy for Breast Cancer.
Acronym: EPOPEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19 SEIN 14
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hormonotherapy; E-monitoring
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with breast cancer treated by adjuvant hormonotherapy (Experimental)
  Interventions: Other: Dedicated and coordinated monitoring

INTERVENTIONS:
Other: Dedicated and coordinated monitoring — * Coordinated monitoring performed by a dedicated nurse: consultation before hormonotherapy initiation
  * Monitoring at home over a period of 6 months using an e-monitoring tool: assessment of adverse events and completion of GIRERD questionnaire at week 3 and week 6.

SUMMARY:
This is a monocentric, prospective cohort study evaluating the feasibility of an E-monitoring protocol in patients with breast cancer treated by adjuvant hormonotherapy .

45 patients will be included.

Patients will be followed during 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient treated for hormone-dependent localized breast cancer with adjuvant HT (tamoxifen or anti-aromatase +/- LHRH agonist)
2. Patient equipped with a computer or tablet computer and an internet connection at home
3. Age > 18 years old
4. Patient affiliated to the french social security system
5. Patient who has signed informed consent before inclusion in the study and before any specific procedures for the study
6. Women of childbearing age should have effective contraception under hormonotherapy

Exclusion Criteria:

1. Patient with breast cancer who does not require adjuvant hormonotherapy
2. Patient with metastatic breast cancer
3. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
4. Patient previously treated for breast cancer (infiltrating or in-situ) with adjuvant HT or not
5. Patient protected by law.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Rate of patients who do not fail the E-Monitoring protocol | 6 months per patient

SECONDARY OUTCOMES:
Number of medical consultations required over 6 months | 6 months per patient
Rate of hormonotherapy adherence evaluated by the GIRERD questionnaire | 6 months per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer Toulouse Oncopole, Toulouse, France